CLINICAL TRIAL: NCT03504826
Title: Walking Rehabilitation After Spinal Cord Injury: Locomotor Training Using Adaptive Robotics
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brooks Rehabilitation (Other)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-02655
Record Dates: First submitted 2018-03-26; First posted 2018-04-20 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injuries
Keywords: adaptive robotics; locomotor training; Spinal Cord diseases; walking rehabilitation; Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Locomotor training using adaptive robot (Experimental): The intervention will consist of 60 sessions of locomotor training using the HAL adaptive robot. The training sessions will be scheduled 5 days per week for 12 weeks. A physical therapist with expertise in SCI walking rehabilitation and use of the HAL will oversee all intervention sessions. The intervention sessions will include up to a total of 40 minutes of stepping time, which may take up to 2 hours to complete due to set up time and rest breaks.
  Interventions: Device: Hybrid Assistive Limb (HAL)

INTERVENTIONS:
Device: Hybrid Assistive Limb (HAL) — Intensive training with the HAL consisting of two components to the intervention session that include: 1) locomotor treadmill training with the HAL device and 2) locomotor training over ground without the HAL device. All training will be overseen by a licensed physical therapist.

SUMMARY:
Locomotor training is an established rehabilitation approach that is beneficial for improving walking function in individuals with spinal cord injuries (SCIs). This approach focuses on repetitive practice and appropriate stepping movements to activate spinal neural networks and promote rhythmic motor output associated with walking. Assistance with stepping movements is often provided by physical therapists and trainers, but this can be costly and difficult to deliver in the cost-constrained U.S. healthcare market. Robotic devices have been used as an alternate method to deliver locomotor training, but current robotic approaches often lack the natural movement variations that characterize normal human stepping. Furthermore, studies to compare locomotor training approaches have not shown any specific benefits of using robotic devices. A new type of robotic device has emerged that uses an individual's muscle activation and stepping movements to control the robot during walking. This adaptive robotic device adjusts to the user's intentions and can assist with stepping during locomotor training in a manner that matches natural human stepping. While this type of adaptive robot has been preliminarily tested, the safety and efficacy of locomotor training using adaptive robotics are not well-established in patients with SCI. This is a critical step to determine if individuals with SCI may benefit from use of this device and for preliminary adoption of this technology. Recent studies have used the Cyberdyne Hybrid Assistive Limb (HAL) to deliver locomotor training and have reported outcomes suggesting that the HAL adaptive robot is safe and efficacious for walking rehabilitation in European SCI patients. Therefore this study will use the HAL adaptive robot to deliver locomotor training. This research is necessary to determine if use of the HAL is potentially beneficial and warranted for use with locomotor training and SCI patients receiving care in the U.S. Results of this study may contribute to the development and implementation of effective walking rehabilitation approaches for people with SCIs.

DETAILED DESCRIPTION:
The purpose of this study is to examine the safety and efficacy of locomotor training using adaptive robotics in adults with chronic SCI. Safety will be determined by monitoring of adverse responses such as skin irritation, pain, changes in spasticity and function. Preliminary efficacy for improving walking function will be determined by tests of walking speed and endurance prior to and following 60 daily sessions of locomotor training using adaptive robots.

Specific Aims:

Specific Aim 1: Test the hypothesis that locomotor training using adaptive robotics such as the Cyberdyne Hybrid Assistive Limb (HAL) is safe for individuals with chronic incomplete spinal cord injury (SCI). Safety will be demonstrated by an adverse response rate that does not exceed the frequency and severity of adverse responses reported for other well-established locomotor rehabilitation approaches. Safety will be assessed by monitoring of specific conditions such as skin integrity, pain, and spasticity.

Specific Aim 2: Test the hypothesis that locomotor training using adaptive robotics such as the Cyberdyne HAL (5x/week for 12 weeks, 60 sessions, 2 hours each) is efficacious for improving walking function in adults with chronic incomplete SCIs. Walking function may be assessed using standard clinical tests to measure walking speed and walking endurance. A battery of clinical tests (listed in Outcome Measures) will be selected for use based on each participant's functional capabilities.

To address the aims of the study, the investigators will use a pre-post repeated measures study design. Following phone and in-person screenings and physician approval, individuals will provide informed consent to the study procedures. Non-invasive tests of physical function and health will be conducted prior to and following 60 sessions of locomotor training using the HAL, an adaptive robotic device that is custom fitted to each individual to provide assistance to the lower limbs during locomotor training.

Subject recruitment: Individuals with chronic SCI (>1 year) who meet the given enrollment criteria (see inclusion and exclusion criteria) will be included for this study. Recruitment will occur from within the Brooks Health System which includes the Brooks Cybernic Treatment Center, as well as from their healthcare providers and advertisements in the community.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 - 80 years old
2. Diagnosed with chronic, sensory or motor incomplete spinal cord injury (ASIA Impairment Scale (AIS) B, C, D), >1 year post injury
3. Medically stable with no acute illness, infections
4. Obtained physician approval to participate in study procedures
5. Able to walk 10 feet with or without assistance, gait assistive devices and/or orthotics
6. Able to provide informed consent

Exclusion Criteria:

1. Additional neurologic conditions such multiple sclerosis, Parkinson's disease, stroke, brain injury
2. Presence of unstable or uncontrolled medical conditions such as cardiovascular disease, myocardial infarction (<1 year), pulmonary infection or illness, renal disease, autonomic dysreflexia, infections, pain, heterotopic ossification
3. Cognitive or communication impairments limiting communication with study staff or ability to provide informed consent
4. Lower extremity joint contractures limiting the ability to stand upright and practice walking
5. Skin lesions or wounds affecting participation in walking rehabilitation
6. Acute or unstable fracture, diagnosis of osteoarthritis or bone impairments affecting safe participation in walking rehabilitation
7. Spasticity or uncontrolled movements limiting participation in walking rehabilitation
8. Body weight or height that is incompatible with safe use of the HAL and/or use of a support harness and body weight support system
9. Pain that limits walking or participation in walking rehabilitation
10. Current participation in rehabilitation to address walking function
11. Botox injections in lower extremity muscles affecting walking function within 4 months of study enrollment
12. Legal blindness or severe visual impairment
13. Known pregnancy
14. Pacemaker or medical device implants which may interfere with the use of the HAL

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
10-Meter Walk Test (10MWT) | Daily and change in baseline to weeks 6 and 12
  Performance assessment of comfortable and fastest safe walking speed for 10 meters. A reduced time (in seconds) to complete the 10-Meter Walk Test reflects improvement in walking function.
6-Minute Walk Test (6MWT) | Daily and change in baseline to weeks 6 and 12
  Performance assessment of walking endurance for 6 minutes. An increase in the number of meters walked during this assessment reflects an improvement in walking endurance.

SECONDARY OUTCOMES:
Electromyogram (EMG) will be used to assess the neuromuscular activation of the lower extremities | Change in baseline to week 12
  A wireless, 16-channel EMG system will be applied at various key muscle groups on both lower extremities. Greater amplitude or changes in activation timing in the EMG signal will reflect improvement in muscle activation.

CONTACTS AND LOCATIONS:
Overall Officials: Emily J Fox, DPT, PhD, Principal Investigator — Brooks Rehabilitation
Locations (1):
- Brooks Rehabilitation, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No